CLINICAL TRIAL: NCT05668468
Title: Can Feeding a Bifido Bacteria That Readily Digests Lactose and Galactooligosacharides Improve Lactose Digestion and Tolerance Through Alteration of the Microbiome?
Brief Title: A Bifido Bacteria to Improve Lactose Digestion and Tolerance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Purdue University (Other)
Responsible Party: Principal Investigator, Dennis A. Savaiano, Professor, Purdue University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: IRB-2021-1099
Record Dates: First submitted 2022-12-07; First posted 2022-12-29 (Actual); Last update posted 2022-12-29 (Actual); Status verified 2022-12

CONDITIONS: Lactose Intolerance
MeSH Terms: conditions — Lactose Intolerance

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: placebo of cellulose identical in size, shape and color to intervention bifidus
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Placebo Comparator): Daily cellulose capsule
  Interventions: Other: Placebo cellulose capsule
- Experimental Group (Experimental): Daily Bifidobacterium adolescentis IVS-1,capsule
  Interventions: Dietary Supplement: Bifidobacterium adolescentis IVS-1 capsule

INTERVENTIONS:
Dietary Supplement: Bifidobacterium adolescentis IVS-1 capsule — Daily Bifidobacterium adolescentis IVS-1 capsule containing up to 6x10 ninth cfu per capsule or daily cellulose capsule
  Arms: Experimental Group
Other: Placebo cellulose capsule — Daily cellulose capsule
  Arms: Control Group

SUMMARY:
We want to determine if feeding a bifido bacteria that readily digests lactose and galactooligosacharides improves lactose digestion and tolerance through alteration of the microbiome.

DETAILED DESCRIPTION:
Bifidobacterium adolescentis IVS-1, is a strain of the bacterial species Bifidobacterium adolescentis that has been thoroughly characterized. It is deposited with the American Type Culture Collection (ATCC®) under Patent Deposit Designation as PTA-120614. B. adolescentis IVS-1 is part of the broader group of bacteria within the genus. These bacteria are one of the major genera of microorganisms that make up the gastrointestinal tract microbiota in mammals. Bifidobacterium is also long considered to contribute to a healthy gastrointestinal tract in infants as well as adults. These organisms have been used in food products and dietary supplements for decades, with a record of safe consumption. B. adolescentis IVS-1 is a specially selected strain. Krumbeck et. al. isolated bifidobacteria from fecal samples of human individuals who had consumed the prebiotic GOS during a previous human trial. For this isolation, a combination of approaches was used to select a candidate strain (B. adolescentis strain IVS-1) enriched by GOS in vivo. The subject consumed increasing doses of GOS for nine weeks. A retrospective analysis of the fecal microbiota of one subject revealed an 8-fold enrichment in B. adolescentis strain IVS-1 during GOS administration. Thus, the strain originated from a subject who showed a strong bifidogenic response to GOS. The functionality of GOS to support the establishment of IVS-1 in the gastrointestinal tract was then evaluated in rats. Strain-specific quantitative real-time PCR showed that the addition of GOS increased B. adolescentis IVS-1 abundance in the distal intestine by nearly two logs. Illumina 16S rRNA sequencing not only confirmed the increased establishment of IVS-1 in the intestine but also revealed that the strain was able to outcompete the resident Bifidobacterium population when provided with GOS. The preparation containing Bifidobacterium adolescentis IVS-1 is manufactured at Centro Sperimentale Del Latte srl, Strada Provinciale per Merlino, 3, 26839, 26839 Zelo Buon Persico LO, Italy, in accordance with current good manufacturing practices (cGMPs); approved and recognized by Global Food Safety Initiative. The facility is FSSC 2200 certified.

Bifidus and lactose intolerance:

The use of probiotics, including Bifidobacterium, has had mixed success in improving lactose tolerance. The failures are likely due to dose and strain, as demonstrated in our lab. Supplementation with Bifidobacterium can change the colonic microflora to improve lactose digestion, and changes in the gut microbiome can mediate lactose intolerance symptoms as first shown in our lab and more recently by others. Bifidobacterium adolescentis IVS-1 presents a unique opportunity to evaluate both species and dose of a very well characterized probiotic in improving lactose digestion, altering the microbiome, and improving lactose tolerance.

Study Procedures:

Participants will undergo a pre-Informed Consent phone screening for eligibility. Informed Consent will be obtained. Demographic/ contact information and a departmental Subject Payment Form will be completed. Study staff contact information and study information handout will be provided. Consented participants will then undergo an abbreviated hydrogen breath test (3 hours duration) which involves drinking 8 oz. of 2% fat commercial milk and giving a breath sample and rating any symptoms they might have at 1 and 2 hours post milk dose. Participants who register a hydrogen value of 20ppm or above will be eligible to proceed to Part 1 of the study.

PART 1: On study:

Days 1-13: Participants will be instructed to avoid lactose intake (i.e. milk in any form, fluid or soft dairy foods, etc.) Participants will be asked to rate any symptoms that are generally associated with lactose intolerance they might be experiencing once daily. This information will be returned daily to study staff electronically, or can be returned to the Clinical Research Center.

Day 11, 12 or 13: Provide a stool sample. Participants can provide this sample on one of the days listed. A range is given to account for participants who may not have a bowel movement daily. Participants will be given a labeled container for stool collection, and return the container to the Clinical Research Center.

Day 14: Eight hour hydrogen Breath Test: Participants will fast for 12 hours prior to the test and the last meal eaten before fasting will be a low fiber meal. Participants will be given food grade lactose in water containing 0.5g lactose per kg body weight (12g per 240ml cup) with a maximum of 50g of lactose. Breath samples will be taken at the following time points: 0 (pre-milk dose), 30 minutes, 60 minutes, 2 hours, 3 hours, 4 hours, 5 hours, 6 hours, 7 hours, and 8 hours for a total of ten (10). Participant will record any symptoms they experience related to lactose intolerance at these same time intervals using provided forms. Participants will be randomized to receive either a daily bifidus capsule (containing up to 5x10 ninth cfu per capsule) or a placebo capsule containing cellulose (Days 15-27).

PART 2: On Study: Days 15-27:

Participants continue to avoid dairy foods. Participants will daily take either a bifidus capsule or a cellulose capsule. Participants will be asked to rate any symptoms that are generally associated with lactose intolerance they might be experiencing once daily.

Day 25, 26, or 27: Provide a stool sample.

Day 28: Eight hour hydrogen breath test:

PART 3: Days 29-43:

Participants will resume their normal diet including dairy foods and will continue to rate symptoms that are associated with lactose intolerance once daily.

Day 40, 41, or 42: Provide a stool sample.

Human subjects recruitment, blinding, and protection:

Staff who interact with subjects will be blinded to treatments. Recruitment efforts include flyers, social media ads, and other local print media. Participant information will be accessible only by study staff. Phone calls will be done in an area allowing for privacy. Research visits will be in the Purdue Clinical Research Center. Risk of breach of confidentiality is possible. Measures will be taken to minimize this risk. Individuals volunteering to participate in this study will be assigned a Subject Identification Number (SID) for data entry and Case Report Form completion. The linking information will be held by the study staff, in a locked file cabinet, in a locked office, and destroyed when the study/publication timeline is completed. Data will be stored both via hard copy and electronically. Hard copies will be stored in a locked file cabinet, in a locked office (Stone Hall, Purdue University, West Lafayette). Electronic data will be maintained in a secure folder, on a secure Purdue server. Only the Principal Investigator and study staff will have access to participant data. Information collected for payment purposes (name, address, social security number) will be provided to the business office, Purdue University for the purpose of facilitating payment. This information will be kept in a locked filing cabinet. No additional identifier will be provided with this information (i.e. Subject Identification Number), so there will be no way of matching this information to their data. All research records and data will be stored for a minimum of 3 years. Records and data will be stored until all analysis/publication activity has ceased.

ELIGIBILITY:
* Inclusion Criteria:

  1. Ability/desire to provide informed consent
  2. Aged 18 to 65 years of age inclusive at screening
  3. Self report of lactose intolerance or lactose maldigestion
  4. Agrees to refrain from all other treatments and products used for dairy intolerance (e.g., Lactaid®, Dietary Supplements, probiotics) during study involvement
  5. Willing to return for all study visits and complete all study related procedures, including fasting before and during the hydrogen breath tests, and avoiding lactose in their diets (ex. milk, fluid, and soft dairy foods) for Days 1-28 of the study
  6. Able to understand and provide written informed consent in English

Exclusion Criteria:

1. Allergic to milk
2. Currently pregnant
3. Currently lactating
4. Cigarette smoking or other use of tobacco or nicotine containing products within 3 months of screening
5. Diagnosed with any of the following disorders known to be associated with abnormal gastrointestinal motility such as; Gastroparesis, amyloidosis, neuromuscular diseases (including Parkinson's disease), collagen vascular diseases, alcoholism, uremia, malnutrition, or untreated hypothyroidism
6. History of surgery that alters the normal function of the gastrointestinal tract including, but not limited to: gastrointestinal bypass surgery, bariatric surgery, gastric banding, vagotomy, fundoplication, pyloroplasty [Note: history of uncomplicated abdominal surgeries such as removal of an appendix more than 12 months prior to screening will not be excluded]
7. Past or present : Organ transplant, chronic pancreatitis, pancreatic insufficiency, symptomatic biliary disease, Celiac disease, chronic constipation, diverticulosis, inflammatory bowel disease (IBD), ulcerative colitis (UC), Crohn's disease (CD), small intestine bacterial overgrowth syndrome (SIBO), gastroparesis, gastro-esophageal reflux disease (GERD), Irritable Bowel Syndrome (IBS) or any other medical condition with symptoms that could confound collection of adverse events.
8. Active ulcers, or history of severe ulcers
9. Diabetes mellitus (type 1 and type 2)
10. Congestive Heart Failure (CHF)
11. Human Immunodeficiency Virus (HIV), Hepatitis B or Hepatitis C
12. BMI > 35 kg/m2
13. Recent bowel preparation for endoscopic or radiologic investigation within four weeks of screening (e.g., colonoscopy prep)
14. Use of concurrent therapy(ies) or other products (e.g., laxatives, stool softeners, Pepto Bismol®,Lactaid® Dietary Supplements, probiotics) used for symptoms of dairy intolerance within 7 days of screening
15. Chronic antacid and/or PPI use
16. Recent use of systemic antibiotics defined as use within 30 days prior to screening
17. Recent high colonic enema, defined as use within 30 days prior to screening
18. Any concurrent disease or symptoms which may interfere with the assessment of the cardinal symptoms of dairy intolerance (i.e., gas, diarrhea, bloating, cramps /stomach pain, fecal urgency)
19. History of ethanol (alcohol) and/or drug abuse in the past 12 months
20. Currently undergoing chemotherapy
21. Use of any investigational drug or participation in any investigational study within 30 days prior to screening
22. Prior enrollment in this study
23. Any other conditions/issues noted by the study staff and/or Principal Investigator that would impact participation and/or protocol compliance

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Bifidus feeding will change lactose digestion | 14 days
  difference in lactose maldigestion as measured by breath hydrogren following a lactose challenges on day 14 and day 28.
Bifidus feeding will change lactose intolerance symptoms | 14 days
  differences in symptoms of flatulence, stomach discomfort, and diarrhea following lactose challenges on day 14 and day 28

SECONDARY OUTCOMES:
daily symptoms of lactose intolerance will be minimal following return to normal diet | 14 days
  daily recording of lactose intolerance symptoms days 29-43 as compared to the control feeding

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Savaiano, PhD, Principal Investigator — Purdue University
Locations (1):
- Purdue University, West Lafayette, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] O'Sullivan MG, Thornton G, O'Sullivan GC, Collins JK. Probiotic bacteria: myth or realilty. Trends in Food Science & Technology. 2010; 3: 309-314
- [Background] Fuller R, Gibson GR. Modification of the intestinal microflora using probiotics and prebiotics. Scand J Gastroenterol Suppl. 1997;222:28-31. doi: 10.1080/00365521.1997.11720714. PMID 9145443
- [Background] Reid G. Safety of lactobacillus strains as probiotic agents. Clin Infect Dis. 2002 Aug 1;35(3):349-50. doi: 10.1086/342477. No abstract available. PMID 12115112
- [Background] Kocian J. Further possibilities in the treatment of lactose intolerance--lactobacilli. Prakticky Lekar. 1994; 74: 212-214.
- [Background] Sharma M, Wasan A, Sharma RK. Recent developments in probiotics: An emphasis on bifidobacterium. Food Bioscience. 2021;41: 100993.
- [Background] Krumbeck JA, Maldonado-Gomez MX, Martinez I, Frese SA, Burkey TE, Rasineni K, Ramer-Tait AE, Harris EN, Hutkins RW, Walter J. In vivo selection to identify bacterial strains with enhanced ecological performance in synbiotic applications. Appl Environ Microbiol. 2015 Apr;81(7):2455-65. doi: 10.1128/AEM.03903-14. Epub 2015 Jan 23. PMID 25616794
- [Background] Davis LM, Martinez I, Walter J, Hutkins R. A dose dependent impact of prebiotic galactooligosaccharides on the intestinal microbiota of healthy adults. Int J Food Microbiol. 2010 Dec 15;144(2):285-92. doi: 10.1016/j.ijfoodmicro.2010.10.007. Epub 2010 Oct 14. PMID 21059476
- [Background] Leis R, de Castro MJ, de Lamas C, Picans R, Couce ML. Effects of Prebiotic and Probiotic Supplementation on Lactase Deficiency and Lactose Intolerance: A Systematic Review of Controlled Trials. Nutrients. 2020 May 20;12(5):1487. doi: 10.3390/nu12051487. PMID 32443748
- [Background] Jiang T, Mustapha A, Savaiano DA. Improvement of lactose digestion in humans by ingestion of unfermented milk containing Bifidobacterium longum. J Dairy Sci. 1996 May;79(5):750-7. doi: 10.3168/jds.S0022-0302(96)76422-6. PMID 8792277
- [Background] He T, Roelofsen H, Alvarez-Llamas G, de Vries M, Venema K, Welling GW, Vonk RJ. Differential analysis of protein expression of Bifidobacterium grown on different carbohydrates. J Microbiol Methods. 2007 May;69(2):364-70. doi: 10.1016/j.mimet.2007.02.008. Epub 2007 Feb 28. PMID 17397953
- [Background] Hertzler SR, Savaiano DA. Colonic adaptation to daily lactose feeding in lactose maldigesters reduces lactose intolerance. Am J Clin Nutr. 1996 Aug;64(2):232-6. doi: 10.1093/ajcn/64.2.232. PMID 8694025
- [Background] Hertzler SR, Savaiano DA, Levitt MD. Fecal hydrogen production and consumption measurements. Response to daily lactose ingestion by lactose maldigesters. Dig Dis Sci. 1997 Feb;42(2):348-53. doi: 10.1023/a:1018822103911. PMID 9052518
- [Background] Brandao Gois MF, Sinha T, Spreckels JE, Vich Vila A, Bolte LA, Weersma RK, Wijmenga C, Fu J, Zhernakova A, Kurilshikov A. Role of the gut microbiome in mediating lactose intolerance symptoms. Gut. 2022 Jan;71(1):215-217. doi: 10.1136/gutjnl-2020-323911. Epub 2021 Mar 18. No abstract available. PMID 34086598
- [Background] Vitellio P, Celano G, Bonfrate L, Gobbetti M, Portincasa P, De Angelis M. Effects of Bifidobacterium longum and Lactobacillus rhamnosus on Gut Microbiota in Patients with Lactose Intolerance and Persisting Functional Gastrointestinal Symptoms: A Randomised, Double-Blind, Cross-Over Study. Nutrients. 2019 Apr 19;11(4):886. doi: 10.3390/nu11040886. PMID 31010241